CLINICAL TRIAL: NCT00956384
Title: Acellular Dermal Matrix in One-Stage Breast Reconstruction: A RCT
Brief Title: One-stage Breast Reconstruction Using Dermal Matrix/Implant Versus Two-stage Expander/Implant Procedure
Acronym: AllodermRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Women's College Hospital (Other); Vancouver General Hospital (Other); Canadian Breast Cancer Foundation (Other); Tom Baker Cancer Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSEF-137034
Record Dates: First submitted 2009-08-07; First posted 2009-08-11 (Estimated); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: Breast reconstruction; Early stage; Skin-saving mastectomy; Prophylactic mastectomy; Acellular dermal matrix; BRCA Mutation Carriers
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Implants; Alloderm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- One-stage dermal matrix/implant (Experimental): One-stage breast reconstruction with dermal matrix and implant
  Interventions: Procedure: One-stage dermal matrix/implant procedure
- Two-stage tissue expander/implant (Active Comparator): Two-stage breast reconstruction with tissue expander and implant
  Interventions: Procedure: Two-stage tissue expander/implant procedure

INTERVENTIONS:
Procedure: One-stage dermal matrix/implant procedure — One-stage breast reconstruction with dermal matrix and implant
  Other Names: Alloderm
  Arms: One-stage dermal matrix/implant
Procedure: Two-stage tissue expander/implant procedure — Two-stage breast reconstruction with tissue expander and implant
  Arms: Two-stage tissue expander/implant

SUMMARY:
Currently the two-stage tissue expander/implant (TE/I) technique is the standard breast reconstructive option for breast cancer patients selected for immediate, skin-sparing mastectomy. This procedure has been demonstrated to be oncologically safe in patients with specific criteria for early stage breast cancer. The primary drawback, however, is that it requires two separate procedures under general anesthesia and multiple office visits for expander inflation to create the breast mound. Acellular dermal matrix has gained widespread acceptance for use in breast reconstruction and other areas and has the potential to provide support to the breast implant without tissue expansion in a one-stage procedure. The purpose of the study is to test this new procedure and to evaluate the impact of one-stage breast reconstruction using acellular dermis compared to the standard two-stage expander/implant technique on measures of patient satisfaction and quality of life.

DETAILED DESCRIPTION:
Recently, there has been significant focus on the performance of skin-sparing mastectomies in certain types of breast cancer patients. These treatments may be performed for prophylactic mastectomy but also have been demonstrated to be oncologically safe in patients with specific criteria for early stage breast cancer. Currently, the two-stage tissue expander/implant (TE/I) technique is the standard breast reconstructive option for breast cancer patients selected for immediate, skin-sparing mastectomy, however there are significant disadvantages as this technique requires two separate surgeries and multiple office visits to complete that may affect a patients quality of life. Medically safe compounds such as acellular dermal matrix have been developed that have the potential to support breast implants without requiring numerous tissue expansions and consequently providing the potential for a one-stage breast implant/reconstruction procedure for immediate, skin-sparing mastectomies.

To examine patient satisfaction, quality of life and overall aesthetic outcome achieved using the acellular dermal matrix facilitated one-staged breast reconstruction at 2 weeks, 6 & 12 months following completion of the reconstruction. Hypothesis 2: Patient satisfaction, quality of life and overall aesthetic outcome achieved using the acellular dermal matrix facilitated one-stage breast reconstruction is superior to that following the standard two-stage tissue expander/ implant breast reconstruction technique in selected mastectomy patients.

To determine the short and long-term operative complication rates associated with the use of dermal matrix in one-stage immediate breast reconstruction following skin-sparing mastectomy. Hypothesis 1: The use of acellular dermal matrix in one-stage immediate prosthetic breast reconstruction is associated with decreased short and long-term postoperative complications compared with the traditional two staged tissue expander/implant procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo immediate, implant-based reconstruction following skin-sparing and nipple-sparing mastectomy.
* Patients who are older than 18 years of age and who understand English enough to complete the study questionnaires.

Exclusion Criteria:

* Patient refusal, patients with documented psychiatric history of psychosis or mental disorder excluding depression, patients who are active smokers.
* Patients who will undergo any of the following: Autologous tissue reconstruction, patients with prior history of radiation or expected to receive post-operative radiation, patients who are pregnant, patients with grade III ptosis.
* Intraoperative exclusion of those whose mastectomy flaps are deemed to be too thin or have significant ischemia.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toni Zhong, MD FRCS(C), Principal Investigator — University Health Network, Toronto; Mitchell Brown, MD FRCS(C), Principal Investigator — Women's College Hospital; Stefan Hofer, MD FRCS(C), Principal Investigator — University Health Network, Toronto; John Semple, MD FRCS(C), Principal Investigator — Women's College Hospital; Brett Beber, MD FRCS(C), Principal Investigator — Women's College Hospital
Locations (4):
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Plastic Surgery, Women's College Hospital, Toronto, Ontario
  - Plastic and Reconstructive Surgery, University Health Network, Toronto, Ontario

REFERENCES:
- [Derived] Zhong T, Temple-Oberle C, Hofer SO, Beber B, Semple J, Brown M, Macadam S, Lennox P, Panzarella T, McCarthy C, Baxter N; MCCAT Study Group. The Multi Centre Canadian Acellular Dermal Matrix Trial (MCCAT): study protocol for a randomized controlled trial in implant-based breast reconstruction. Trials. 2013 Oct 28;14:356. doi: 10.1186/1745-6215-14-356. PMID 24165392

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | One-stage Dermal Matrix/Implant | Two-stage Tissue Expander/Implant
Started | 102 | 96
Completed | 86 | 78
Not Completed | 16 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | One-stage Dermal Matrix/Implant | Two-stage Tissue Expander/Implant | Total
Number analyzed (Participants) | 86 | 78 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 86 | 78 | 164
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.9 (8.4) | 46 (11.2) | 45.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 78 | 164
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 20 | 7 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 6 | 14
  White | 58 | 65 | 123
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 86 | 78 | 164

OUTCOME MEASURES:

1. Primary Outcome: BreastQ Quality of Life and Satisfaction Questionnaire
Description: Compare the change in the patient satisfaction and QOL scores between one-stage ADM-assisted and two-stage TE/I reconstruction without ADM over time (at 2 weeks after mastectomy, at 6 months and at 12 months following the final reconstruction procedure) from baseline scores following reconstruction using the validated BREAST-Q reconstruction module.
  The BREAST-Q Reconstruction Module is used to measure outcomes across four domains/sub-scales: satisfaction with the breast, psychosocial wellbeing, physical wellbeing, and sexual wellbeing. Each domain is scored on a scale of 1 to 100, with higher scores indicating better quality of life and greater patient satisfaction with more favorable outcomes.
Time Frame: 12 months post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | One-stage Dermal Matrix/Implant | Two-stage Tissue Expander/Implant
Number analyzed (Participants) | 86 | 78
score on a scale | 65.32 (13.63) | 67.07 (16.05)
Statistical Analysis 1: Comparison: One-stage Dermal Matrix/Implant vs Two-stage Tissue Expander/Implant; For the comparison of mean BREAST-Q subdomain score at each timepoint, Mann-Whitney U test was used for skewed data, while independent t-test was used for not skewed data. We investigated the possibly variable effects of the treatment group differences across multiple time-points, namely 2 weeks after mastectomy, at 6 months and at 12 months following the reconstruction procedure. A linear regression model was used to account for the correlation between the three time-points within each patient; Test type: Superiority — A minimally clinically important difference of 4 as statistically significant at the 0.05 level (two-sided), with a power equal to 0.85; p = 0.05, t-test, 2 sided — Threshold for statistical significance was p= 0.05; Mean Difference (Final Values) = -2.69, 95% CI 2-sided [-10.57 to 5.19]

2. Secondary Outcome: Number of Participants With Short Term Surgical Complications
Description: Short complication rates were collected prospectively on intraoperative and postoperative assessment forms. Short-term complications were those that occur intraoperatively or within the first 2 months of surgery
Time Frame: 6- months post-op
Measure: Count of Participants; unit: Participants
Arm/Group | One-stage Dermal Matrix/Implant | Two-stage Tissue Expander/Implant
Number analyzed (Participants) | 86 | 78
Participants | 32 | 27
Statistical Analysis 1: Comparison: One-stage Dermal Matrix/Implant vs Two-stage Tissue Expander/Implant; We assessed the effect of the surgical method on the occurrences of any complications versus none via logistic regression, and results were expressed as odds ratios with 95% CIs; Test type: Superiority; p < 0.05, Regression, Logistic

3. Secondary Outcome: Number of Participants With Long Term Surgical Complications
Description: Long-term minor and major surgical complication rates were documented and collected prospectively on intraoperative and postoperative assessment form at 12-months follow-up visit
Time Frame: 12 months post-op
Measure: Count of Participants; unit: Participants
Arm/Group | One-stage Dermal Matrix/Implant | Two-stage Tissue Expander/Implant
Number analyzed (Participants) | 86 | 78
Participants | 23 | 12

ADVERSE EVENTS:
Time Frame: 2 years
Description: Chart reviewed on a regular schedule.
Arm/Group | One-stage Dermal Matrix/Implant | Two-stage Tissue Expander/Implant
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/78
Other Adverse Events (participants affected / at risk) | 7/86 | 6/78
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | One-stage Dermal Matrix/Implant (N=86) | Two-stage Tissue Expander/Implant (N=78)
Implant or TE exposure (Surgical and medical procedures) | 7 (7) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-06-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT00956384/Prot_SAP_000.pdf